CLINICAL TRIAL: NCT07384728
Title: The Impact of Ramadan Experiences on Treatment, Psychological and Glycemic Control Levels, and Adherence in Individuals With Type 2 Diabetes
Brief Title: Ramadan Experience of Individuals With Type 2 Diabetes
Acronym: Randomized
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dilan aktepe coşar (Other)
Collaborators: Gümüşhane Universıty (Other)
Responsible Party: Sponsor-Investigator, Dilan aktepe coşar, lecture, Gümüşhane Universıty
Organization: Gümüşhane Universıty (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hm20260001
Record Dates: First submitted 2026-01-06; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Ramadan experience; Treatment; Psychological; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This research is a clinical trial designed to examine the effects of fasting during Ramadan on treatment adherence, psychological adjustment, and glycemic control in individuals with type 2 diabetes. The study compares individuals who fast and those who do not fast during Ramadan to evaluate the relevant variables. Participants are monitored before and after Ramadan; glycemic control, treatment adherence, and psychological adjustment are measured using standardized measurement tools. The study model aims to guide clinical practice and nursing care with the results obtained.
Masking Description: Patients were randomly assigned to groups, and interviews were scheduled at different times to minimize the possibility of interaction between them. Additionally, patients were informed about the study and their consent was obtained prior to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Individuals observing the fast. (Experimental): Patients in the experimental group received face-to-face dietary education from the researcher in the waiting room for approximately 15 minutes, and were given an "Information Brochure." Pre-education (pre-test) data collection tools were administered to diabetic patients. All data collection tools were administered to these patients, except for the structured Patient Information Form, which was completed one month after Ramadan 2026.
  Interventions: Other: The effect of fasting and not fasting during Ramadan.
- No Intervention: Control Group (No Intervention): Diabetic patients in this group were classified as a non-fasting group. No intervention was applied. Only data collection forms were administered before the study (pre-test) and after Ramadan 2026.

INTERVENTIONS:
Other: The effect of fasting and not fasting during Ramadan. — The effects of fasting and non-fasting during Ramadan on treatment adherence, psychological adjustment, and glycemic control.
  Other Names: The effect of fasting during Ramadan
  Arms: Experimental group: Individuals observing the fast.

SUMMARY:
This study aims to examine the effects of fasting during Ramadan on treatment adherence, psychological adjustment, and glycemic control in individuals with type 2 diabetes. While Ramadan fasting is a religious practice, it can also pose health risks such as hypoglycemia, hyperglycemia, and metabolic imbalance in individuals with diabetes. Adherence to treatment and self-care, as well as psychosocial adjustment, are crucial in the effective management of diabetes. Given that a large portion of Turkey's population is Muslim, comparing individuals with type 2 diabetes who fast and those who do not during Ramadan will contribute to improving patient care within a cultural and religious context. The findings of this study are expected to guide nurses in developing personalized, culturally sensitive care plans tailored to the needs of individuals before, during, and after Ramadan.

DETAILED DESCRIPTION:
Fasting during Ramadan is a religious practice observed globally by adult Muslims. Individuals fast during Ramadan due to an emotional and spiritual connection to the holy month. Fasting involves abstaining from food, drink, and oral medications for a month, between sunrise and sunset each year. The duration of Ramadan fasting varies between 10 and 19 hours depending on geographical and seasonal conditions. While this is a religious practice, those who fast may experience various health risks, particularly for individuals with type 1 and type 2 diabetes.

Diabetes mellitus is an insidious chronic metabolic disease characterized by high blood sugar levels that cause serious damage to all body systems over time. Diabetes is a chronic disease that has increased in recent years and leads to morbidity, loss of productivity, decreased quality of life, and mortality in individuals due to various complications. Adherence to treatment plays a critical role in the treatment, care, and management of chronic diseases.

According to the WHO, adherence to treatment in diabetic patients is defined as a self-care process that includes home blood sugar monitoring, regulation of food consumption, medication use, regular physical activity, foot care, regular visits to the doctor for periodic check-ups, and dental care. Individuals who adhere to treatment in chronic diseases can exhibit effective coping skills, avoid psychological problems, experience fewer negative emotions, implement healthy lifestyle changes, and maintain control over their health status.

The psychological aspect of chronic diseases is often underestimated. Although it is assumed that most patients adapt well to the psychological aspects of chronic diseases, it becomes more difficult to adapt psychologically when patients experience deficiencies in their physical health status. Diabetes is a chronic disease that leads to mental and cognitive problems in addition to physiological complications, and it takes time to cope with it. Therefore, understanding the psychosocial adaptation to the disease in individuals with diabetes will guide nurses in positively influencing disease management and preventing or delaying possible complications. In addition, fasting negatively affects individuals with diabetes physically, socially, and psychologically. Glycemic control before Ramadan is considered a key determinant of fasting safety in individuals with diabetes.

In light of this information, and given that the Turkish population is predominantly Muslim, this study aims to examine the effects of fasting and non-fasting during Ramadan on treatment adherence, psychological adjustment, and glycemic control in individuals with Type 2 diabetes. The results of this study are expected to guide healthcare professionals, particularly nurses who have the most contact with patients, in understanding cultural and religious practices before, during, and after Ramadan to provide personalized care tailored to patients' needs. Through this study, we aimed to identify effective strategies to improve both treatment adherence and psychological adjustment by positively impacting the treatment, care, and management of diabetic patients

ELIGIBILITY:
Inclusion Criteria:

Individuals ≥18 years of age

Able to give informed consent

Diagnosed with type 2 diabetes

Planning to fast during Ramadan

Exclusion Criteria:

Presence of psychiatric illness

Presence of cognitive impairment

Receiving additional treatments that significantly affect glucose levels (e.g., ongoing steroid therapy)

Individuals who have decided not to fast during Ramadan

Individuals who have stopped fasting during Ramadan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
1. Parametre | 2-4 weeks
  HbA1c 2-4 weeks before Ramadan (basic assessment).
2. Parametre | 2-4 weeks
  Treatment Adherence Scale, 2-4 weeks before Ramadan This scale was developed to evaluate "Patient Adherence in Type 2 Diabetes Mellitus Treatment." Validity and reliability analyses have shown it to be a valid and reliable scale. Based on the scores obtained from the scale, adherence is considered good if patients are doing what they should and not doing what they shouldn't, despite factors affecting treatment adherence.
  The scale:
  * Is administered to patients with type 2 diabetes for at least one year. • Consists of 30 items in total.
  * A 5-point Likert scale is used for scoring. • Patients indicate the most appropriate option for each statement on the scale using a 5-point Likert scale (Strongly agree=1, Agree=2, Partially agree=3, Disagree=4, and Strongly disagree=5). • The scale contains 13 items representing positive attitudes and 17 items representing negative attitudes. In scoring, positive items (1, 3, 5, 8, 13, 15, 16, 17, 19, 23, 25, 26, 29) are scor
3. Parametre | 2-4 weeks
  Psychological and Adherence Impact Scale 2-4 weeks before Ramadan. The BASE-6 was developed by Cruz et al. (2019) and it is a self-report instrument of general psychological adjustment comprising of six items. Each item assesses how a participant has been feeling in the past week. Items are rated on a 7-point scale (ranging from 1 = Not at all to 5 = Extremely).
  A sample item is "To what extent have you felt irritable, angry, and/or resentful this week?". Using three different adult samples, the original study demonstrated good internal consistency (α = .87-.93) and test-retest reliability (intraclass correlation was .77) over one-week period.
Post-Ramadan 2. Parametre | Post-Ramadan: 1-2 months after
  Treatment adherence will be assessed using the Treatment Adherence Scale for Type 2 Diabetes Mellitus, a validated and reliable 30-item, 5-point Likert scale. Patients rate each item from strongly agree to strongly disagree. Higher scores indicate better adherence to diabetes treatment.

SECONDARY OUTCOMES:
Post-Ramadan 1. Parametre | Post-Ramadan: 1-2 months after
  Post-Ramadan: 1-2 months after the end of fasting (follow-up). Measurements: HbA1c
Post-Ramadan 3. Parametre | Post-Ramadan: 1-2 months after
  Post-Ramadan: 1-2 months after the end of fasting (follow-up). Measurements: The BASE-6 was developed by Cruz et al. (2019) and it is a self-report instrument of general psychological adjustment comprising of six items. Each item assesses how a participant has been feeling in the past week. Items are rated on a 7-point scale (ranging from 1 = Not at all to 5 = Extremely).
  A sample item is "To what extent have you felt irritable, angry, and/or resentful this week?". Using three different adult samples, the original study demonstrated good internal consistency (α = .87-.93) and test-retest reliability (intraclass correlation was .77) over one-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Dilan aktepe coşar, PhD, Study Director — Gümüşhane Universıty
Locations (2):
- Turkey (Türkiye) (2):
  - Gümüşhane Universıty, Gümüşhane, Kelkit
  - Gümüşhane Üniversitesi, Gümüşhane, Kelkit

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared due to the need to protect participant confidentiality, the privacy of personal health information, and compliance with applicable ethical committee approval and data protection legislation (KVKK). Data will only be analyzed for scientific purposes in an anonymized and aggregated form, and there are no plans to share raw data containing individually identifying information with third parties. This approach has been adopted to protect participant rights and ensure compliance with ethical research principles.